CLINICAL TRIAL: NCT07237321
Title: Peripheral Magnetic Stimulation of Foot Muscles
Brief Title: Peripheral Magnetic Stimulation of Foot Muscles: Effects on Medial Longitudinal Arch Height and Foot Muscle Strength in Adults With Flat Feet
Acronym: rPMS-Foot
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Ljubljana (Other)
Collaborators: University of Ljubljana, Faculty of Medicine (Other)
Responsible Party: Principal Investigator, Ales Dolenec, Associate Professor, Faculty of Sport, University of Ljubljana, University of Ljubljana
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: rPMS, 0124-0043; P5-0124, P3-0043 (Other: Slovenian Research and Innovation Agency (ARIS))
Record Dates: First submitted 2025-11-14; First posted 2025-11-19 (Actual); Last update posted 2025-11-25 (Actual); Status verified 2025-11

CONDITIONS: Pes Planus; Flatfoot; Posterior Tibial Tendon Dysfunction
Keywords: Medial Longitudinal Arch; Flatfoot; rPMS; foot invertors; tibialis posterior; repetitive peripheral magnetic stimulation; foot; posterior tibial tendon dysfunction; strength; ultrasound; muscle cross-sectional area
MeSH Terms: conditions — Flatfoot; Posterior Tibial Tendon Dysfunction

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The radiologist and the investigator responsible for testing the strength of the foot invertor muscles will be blinded to group allocation and intervention status. The radiologist will perform all ultrasound assessments of the foot invertor muscles and the height of the medial longitudinal arch, while the investigator will conduct standardized isometric strength measurements of the subtalar joint invertor muscles using a custom isometric dynamometer designed to measure torque along the subtalar axis. Both assessors will remain unaware of whether participants receive active rPMS or no stimulation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rPMS Stimulation Group (Experimental): Subjects in this group will receive repetitive peripheral magnetic stimulation (rPMS) of the foot invertor muscles three times per week for 12 weeks. Stimulation will be applied to the upper third of the anteromedial side of the shin. Intrinsic foot muscles will be simultaneously stimulated using a foot stimulator, with the nondominant foot placed on the stimulation platform. Participants in the experimental group will complete ultrasound imaging, navicular drop assessment, clinical evaluation of the plantar arch index, and isometric strength testing of the foot invertor muscles at three time points: before the intervention (baseline), after 6 weeks, and after 12-week stimulation period.
  Interventions: Device: Repetitive Peripheral Magnetic Stimulation (rPMS)
- Control Group (no stimulation) (No Intervention): Subjects in control group will not receive any stimulation but will undergo the same measurement procedures as the experimental group, including ultrasound imaging, navicular drop assessment, clinical evaluation of the plantar arch index, and isometric strength testing of the foot invertor muscles before and after the 6- and 12-week period.

INTERVENTIONS:
Device: Repetitive Peripheral Magnetic Stimulation (rPMS) — Repetitive peripheral magnetic stimulation (rPMS) will be applied to the foot invertor muscles three times per week for 12 weeks. Stimulation will target the upper third of the anteromedial side of the shin, near the tibia, using an oval magnetic coil. To ensure correct coil placement, visible muscle contraction and ankle inversion will be monitored. Intrinsic foot muscles will be simultaneously stimulated using a foot stimulator, with the nondominant foot positioned on the stimulation platform. Participants will perform isometric inversion contractions during rPMS to enhance neuromuscular activation and short-foot exercises to engage local foot stabilizers.
  Other Names: Peripheral Magnetic Stimulation; rPMS; FMS; Functional Magnetic Stimulation
  Arms: rPMS Stimulation Group

SUMMARY:
This study examines the effects of repetitive peripheral magnetic stimulation (rPMS) on foot invertor muscle strength, morphology, and the height of the medial longitudinal arch (MLA) in individuals with flat feet. The rPMS will be applied non-invasively to the extrinsic and intrinsic foot muscles three times per week for twelve weeks. The experimental group will receive rPMS targeting the invertor muscles of the foot, while the control group will not receive stimulation but will follow the same measurement schedule.

Assessments will be performed at baseline, after 6 weeks, and after 12 weeks of intervention. The primary outcome will be the change in the height of the MLA, evaluated using dynamic navicular drop assessment during gait. Secondary outcomes will include changes in the isometric inversion torque of the foot invertors and morphological adaptations of the tibialis posterior muscle assessed by ultrasound imaging.

This study seeks to determine whether rPMS can improve the height of the MLA, foot invertor muscle strength and structural stability in adults with flat feet. The findings may contribute to developing new, non-invasive therapeutic approaches for improving foot function and preventing musculoskeletal imbalances related to flat foot deformity.

DETAILED DESCRIPTION:
During movement, the role of the foot muscles is often overlooked. Through their strength and stabilizing function, foot muscles play an important role in maintaining balance, posture, and force transmission throughout the body. Proper activation of these muscles also helps preserve the stability of the medial longitudinal arch (MLA), thereby influencing the overall biomechanics of human movement.

The foot muscles are classified as extrinsic (originating outside the foot) and intrinsic (originating and inserting within the foot). Extrinsic muscles, primarily stabilize the ankle joint and control larger movements, whereas intrinsic muscles store and release elastic energy within the foot, contributing to arch support and movement efficiency.

A lowered height or collapsed arch of the foot, known as flat foot (pes planus), is characterized by arch flattening during weight-bearing and affects approximately 13-27% of the adult population. This deformity alters force distribution and shock absorption, increasing mechanical load on the joints and muscles of the lower kinetic chain. Consequently, flat feet are often associated with foot pain, tendinopathies, and different musculoskeletal disorders in the knees, hips, and lumbar spine.

One of the main causes of flat foot deformity is dysfunction of the tibialis posterior (TP) tendon. This dysfunction leads to reduced muscle strength, decreased neuromuscular activation of the foot invertors and plantar flexors, and subsequent lowering of the navicular bone, resulting in a reduced MLA height. Strengthening the m. TP not only maintains arch position but also improves gait efficiency by reducing compensatory activation of other muscles. This muscle is considered as the strongest foot invertor and has the largest moment arm along the subtalar axis.

Recent research highlights that strengthening foot invertor muscles, particularly m. TP, can effectively increase height of the MLA. Conventional interventions include specific exercise programs and proprioceptive neuromuscular facilitation techniques. However, neuromuscular electrical stimulation used in previous studies did not showed significant increases in MLA height, partly due to pain and discomfort during deep muscle stimulation.

Repetitive peripheral magnetic stimulation (rPMS) has emerged as a promising non-invasively alternative, capable of stimulating deep neuromuscular structures. Several studies have shown that high-frequency rPMS can induce muscle activation, transient swelling, and potential hypertrophy indicators. Nevertheless, there is limited evidence on the long-term (multi-week) effects of rPMS on deep muscles such as the m. TP.

Aim of this research is to implement a 12-week rPMS protocol targeting both extrinsic and intrinsic foot invertor muscles, and to examine whether rPMS induces changes in the height of the MLA. Additionally, the study aims to determine whether 12-week rPMS protocol contributed to increased strength and cross-sectional area of the m. TP.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 50 years,
* functionally flat feet of participants.

Exclusion Criteria:

* Acute leg injuries,
* diabetes,
* vascular disorders of the lower limbs,
* open wounds or skin lesions on the lower leg or foot,
* participants with metal implants near the stimulation site,
* cardiac pacemaker,
* other orthopedic or neurological conditions that could affect the study results or pose a health risk to the participants.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12-15 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Change in medial longitudinal arch height | Baseline (Day 1), Week 6, Week 12
  Measuring dynamic navicular drop assessment during the stance phase of gait.

SECONDARY OUTCOMES:
Change in isometric inversion torque of the stimulated foot | Baseline (Day 1), Week 6, Week 12
  Measured using an special designed isometric device to assess maximal voluntary torque during foot inversion in subtalar exis.

OTHER OUTCOMES:
Change in cross-sectional area of the tibialis posterior muscle | Baseline (Day 1), Week 6, Week 12
  Measured using ultrasound imaging to evaluate morphological adaptations of the tibialis posterior muscle and/or other foot invertor muscles.

CONTACTS AND LOCATIONS:
Overall Officials: Rok Bavdek, PhD, Principal Investigator; Nejc Umek, MD PhD, Study Director — Institute of Anatomy, Faculty of Medicine, University of Ljubljana; Jure Jelenc, PhD, Study Director — Iskra Medical, d.o.o.
Locations (1):
- Faculty of Sport, University of Ljubljana, Ljubljana, Ljubljana, Slovenia

IPD SHARING:
Plan to Share IPD: Yes
All de-identified IPD (demographics, primary and secondary outcome measures) will be shared.
Supporting Information: Study Protocol
Time Frame: IPD will be available 12 months after publication of the results and will remain available for 5 years.
Access Criteria: Researchers will be able to request access to IPD. Access will be granted upon reasonable proposals which will be reviewed and approved by the study investigators. Only de-identified datasets will be shared. Data will be provided electronically.
URL: https://www.fsp.uni-lj.si

REFERENCES:
- [Result] Zschorlich V, Yamaguchi T, Schneider C. Editorial: The use of repetitive peripheral magnetic stimulation (rPMS) in neurological disorders and neurorehabilitation. Front Neurol. 2023 Nov 20;14:1324882. doi: 10.3389/fneur.2023.1324882. eCollection 2023. No abstract available. PMID 38053798
- [Result] Hirono T, Ikezoe T, Taniguchi M, Nojiri S, Tanaka H, Ichihashi N. Acute effects of repetitive peripheral magnetic stimulation following low-intensity isometric exercise on muscle swelling for selective muscle in healthy young men. Electromagn Biol Med. 2021 Jul 3;40(3):420-427. doi: 10.1080/15368378.2021.1907402. Epub 2021 Mar 25. PMID 33764250
- [Result] Masse-Alarie H, Flamand VH, Moffet H, Schneider C. Peripheral neurostimulation and specific motor training of deep abdominal muscles improve posturomotor control in chronic low back pain. Clin J Pain. 2013 Sep;29(9):814-23. doi: 10.1097/AJP.0b013e318276a058. PMID 23370067
- [Result] Neugebauer R. [Surgical treatment of colon cancer. 4. Preoperative preparation of the colon]. Aktuelle Probl Chir Orthop. 1979;(10):38-40. No abstract available. German. PMID 32789
- [Result] Baek J, Park N, Lee B, Jee S, Yang S, Kang S. Effects of Repetitive Peripheral Magnetic Stimulation Over Vastus Lateralis in Patients After Hip Replacement Surgery. Ann Rehabil Med. 2018 Feb;42(1):67-75. doi: 10.5535/arm.2018.42.1.67. Epub 2018 Feb 28. PMID 29560326
- [Result] Yang SS, Jee S, Hwang SL, Sohn MK. Strengthening of Quadriceps by Neuromuscular Magnetic Stimulation in Healthy Subjects. PM R. 2017 Aug;9(8):767-773. doi: 10.1016/j.pmrj.2016.12.002. Epub 2017 Jan 8. PMID 28082179
- [Result] Aenumulapalli A, Kulkarni MM, Gandotra AR. Prevalence of Flexible Flat Foot in Adults: A Cross-sectional Study. J Clin Diagn Res. 2017 Jun;11(6):AC17-AC20. doi: 10.7860/JCDR/2017/26566.10059. Epub 2017 Jun 1. PMID 28764143
- [Result] Kelly LA, Farris DJ, Cresswell AG, Lichtwark GA. Intrinsic foot muscles contribute to elastic energy storage and return in the human foot. J Appl Physiol (1985). 2019 Jan 1;126(1):231-238. doi: 10.1152/japplphysiol.00736.2018. Epub 2018 Nov 21. PMID 30462568
- [Result] Beaulieu LD, Schneider C. Repetitive peripheral magnetic stimulation to reduce pain or improve sensorimotor impairments: A literature review on parameters of application and afferents recruitment. Neurophysiol Clin. 2015 Sep;45(3):223-37. doi: 10.1016/j.neucli.2015.08.002. Epub 2015 Sep 9. PMID 26363684
- [Result] Ross MH, Smith MD, Mellor R, Vicenzino B. Exercise for posterior tibial tendon dysfunction: a systematic review of randomised clinical trials and clinical guidelines. BMJ Open Sport Exerc Med. 2018 Sep 19;4(1):e000430. doi: 10.1136/bmjsem-2018-000430. eCollection 2018. PMID 30271611
- [Result] Kohls-Gatzoulis J, Angel JC, Singh D, Haddad F, Livingstone J, Berry G. Tibialis posterior dysfunction: a common and treatable cause of adult acquired flatfoot. BMJ. 2004 Dec 4;329(7478):1328-33. doi: 10.1136/bmj.329.7478.1328. No abstract available. PMID 15576744
- [Result] Jia Y, Sai X, Zhang E. Comparing the efficacy of exercise therapy on adult flexible flatfoot individuals through a network meta-analysis of randomized controlled trials. Sci Rep. 2024 Sep 11;14(1):21186. doi: 10.1038/s41598-024-72149-w. PMID 39261538
- [Result] Hegazy F, Aboelnasr E, Abuzaid M, Kim IJ, Salem Y. Comparing Validity and Diagnostic Accuracy of Clarke's Angle and Foot Posture Index-6 to Determine Flexible Flatfoot in Adolescents: A Cross-Sectional Investigation. J Multidiscip Healthc. 2021 Sep 27;14:2705-2717. doi: 10.2147/JMDH.S317439. eCollection 2021. PMID 34611407
- [Result] Michaudet C, Edenfield KM, Nicolette GW, Carek PJ. Foot and Ankle Conditions: Pes Planus. FP Essent. 2018 Feb;465:18-23. PMID 29381041
- [Result] Dowling GJ, Murley GS, Munteanu SE, Smith MM, Neal BS, Griffiths IB, Barton CJ, Collins NJ. Dynamic foot function as a risk factor for lower limb overuse injury: a systematic review. J Foot Ankle Res. 2014 Dec 19;7(1):53. doi: 10.1186/s13047-014-0053-6. eCollection 2014. PMID 25598843
- [Result] de Souza TMM, de Oliveira Coutinho VG, Tessutti VD, de Oliveira NRC, Yi LC. Effects of intrinsic foot muscle strengthening on the medial longitudinal arch mobility and function: A systematic review. J Bodyw Mov Ther. 2023 Oct;36:89-99. doi: 10.1016/j.jbmt.2023.05.010. Epub 2023 Jun 10. PMID 37949605
- [Result] Johnson AW, Bruening DA, Violette VA, Perkins KV, Thompson CL, Ridge ST. Ultrasound Imaging Is Reliable for Tibialis Posterior Size Measurements. J Ultrasound Med. 2020 Dec;39(12):2305-2312. doi: 10.1002/jum.15340. Epub 2020 May 15. PMID 32412115